CLINICAL TRIAL: NCT05148117
Title: Mitochondrial Dysfunction Contributes to Sepsis Induced Cardiac Dysfunction
Status: Not yet recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Riaz Karukappadath, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: 300007609
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- suspected sepsis group: We will perform a prospective observational study of patients admitted to the intensive care units (ICU) with suspected sepsis or septic shock.
  Interventions: Diagnostic Test: Suspected Sepsis Group - Diagnostic Measurements
- control group: This group will be compared to suspected sepsis or sepsis shock patients. The control group will be age matched, gender-matched, and cardiovascular risk-factor matched controls.
  Interventions: Diagnostic Test: Control Group - Diagnostic Measurements

INTERVENTIONS:
Diagnostic Test: Suspected Sepsis Group - Diagnostic Measurements — Blood samples (7.5ml) will be collected in cell free DNA collection tubes cfDNA will be extracted with the use of MagMAX cell free DNA isolation kit. Quantitative PCR will determine the total cfDNA. cfDNA (5micro litr) will be subjected to bisulphide conversion with use of EZ DNA methylation kit (Zymo research). We will perform digital PCR for interrogating bisulphide treated cfDNA for FMA 101A locus with the use of Quant Studio 3D digital PCR system. Copy numbers of unmethylated FAM 101A locus as determined by d PCR in the sample will be expressed as the copy numbers of cardiomyocyte specific cfDNA per plasma volume.Inflammatory markers IL-6.IL-8, IL 1-18 and C-reactive protein (CRP) will be measured using commercial assays. Speckle tracking imaging will be used to obtain tissue displacement, velocity, strain, and strain rate in radial longitudinal and circumferential planes EF and FS will be determined by conventional methods.
  Groups: suspected sepsis group
Diagnostic Test: Control Group - Diagnostic Measurements — Blood samples (7.5ml) will be collected in cell free DNA collection tubes cfDNA will be extracted with the use of MagMAX cell free DNA isolation kit. Quantitative PCR will determine the total cfDNA. cfDNA (5micro litr) will be subjected to bisulphide conversion with use of EZ DNA methylation kit (Zymo research). We will perform digital PCR for interrogating bisulphide treated cfDNA for FMA 101A locus with the use of Quant Studio 3D digital PCR system. Copy numbers of unmethylated FAM 101A locus as determined by d PCR in the sample will be expressed as the copy numbers of cardiomyocyte specific cfDNA per plasma volume.Inflammatory markers IL-6.IL-8, IL 1-18 and C-reactive protein (CRP) will be measured using commercial assays. Speckle tracking imaging will be used to obtain tissue displacement, velocity, strain, and strain rate in radial longitudinal and circumferential planes EF and FS will be determined by conventional methods.
  Groups: control group

SUMMARY:
This proposal hypothesizes that mitochondrial bioenergetics in the patient will correspond to mtDNA DAMPs levels and markers of inflammation. We predict these will serve as a prognostic indicator of Sepsis induced cardiac dysfunction (SICD) outcomes. Successful completion of these studies will provide a clearer understanding of the etiology of SICD development and therefore will have a high impact on biomedical research by identifying a new mechanism for understanding sepsis induced organ failure. Importantly, they will also provide a means for more directed and focused therapies, based upon individual bioenergetic/mitochondrial-mediated inflammation profiles. The combined, complementary expertise of the Mentor/co-primary investigators (Drs. Mathru and Ballinger) provide an excellent combination in both basic and translational research. They also have experience conducting studies and publications that will strengthen this research project. Importantly, the methods for characterizing mitochondrial bioenergetics from platelets were developed here at UAB, and methods for quantitative assessment of mtDNA DAMPs have been recently developed.

DETAILED DESCRIPTION:
Sepsis induced cardiac dysfunction (SICD) occurs in ~ 50% of the patients with severe sepsis and septic shock, with significant implications for patient's survival. Currently, the precise pathophysiological mechanisms leading to cardiac dysfunction are not fully understood, nor is there an effective therapy for SICD except antibiotics, source control and restoration of hemodynamics to improve organ perfusion.

SICD is characterized by minimal cell death, normal coronary perfusion, preserved tissue oxygen tension and reversibility in survivors. These characteristics point toward an oxygen utilization problem due to mitochondrial dysfunction; interestingly, sepsis mouse models demonstrated an improvement in cardiac function and decreased mortality when they were treated with mitochondrial targeted therapies, consistent with a growing body of evidence that suggests dysregulated mitochondrial metabolism plays a pivotal role in the pathogenesis of SICD. Ultrastructural and functional abnormalities of mitochondria have also been demonstrated in early sepsis, and reactive oxygen species (ROS) generated from mitochondria along with calcium overload trigger mitochondrial permeability transition pore (mPTP) opening which facilitates the externalization of mitochondrial DNA (mtDNA) fragments. These mtDNA fragments, or mtDNA Damage Associated Molecular Patterns (mtDNA DAMPs), activate innate immune response pathways - these pathways are well known to be significant components of intramyocardial inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years old
* With clinical symptoms suggestive of sepsis Control Group
* age matched
* gender matched
* cardiovascular risk factor matched

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study patients admitted to the intensive care unit with suspected sepsis shock will be enrolled and compared to the control group.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2025-12-07 (Estimated); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial dysfunction characterized by bioenergetic changes | within 6 hours of admission to the ICU
  that mitochondrial dysfunction, characterized by bioenergetic changes (dysfunction) is associated with sepsis in humans, and will be significantly linked with mtDNA DAMPs levels and inflammatory markers in the pathophysiology of SICD.
Mitochondrial dysfunction characterized by bioenergetic changes | within 72 hours post admission
  that mitochondrial dysfunction, characterized by bioenergetic changes (dysfunction) is associated with sepsis in humans, and will be significantly linked with mtDNA DAMPs levels and inflammatory markers in the pathophysiology of SICD.
Mitochondrial dysfunction characterized by bioenergetic changes | after clinical recovery from sepsis (approximately 1 month)
  that mitochondrial dysfunction, characterized by bioenergetic changes (dysfunction) is associated with sepsis in humans, and will be significantly linked with mtDNA DAMPs levels and inflammatory markers in the pathophysiology of SICD.
Mitochondrial function in heart | within 6 hours of admission to the ICU
  changes in mitochondrial bioenergetics associated with sepsis can result in differential releases of mtDNA DAMPs, which contribute in inflammation
Mitochondrial function in heart | within 72 hours post admission
  changes in mitochondrial bioenergetics associated with sepsis can result in differential releases of mtDNA DAMPs, which contribute in inflammation
Mitochondrial function in heart | after clinical recovery from sepsis (approximately 1 month)
  changes in mitochondrial bioenergetics associated with sepsis can result in differential releases of mtDNA DAMPs, which contribute in inflammation
Mitochondria and SICD | within 6 hours of admission to the ICU
  examining the potential roles for increased reactive oxygen species (ROS) and nitric oxide (NO) production in SICD using mouse models of sepsis have shown that genetic and/or pharmacologic manipulation of these species decreased oxidative stress, increased ATP generation and restored cardiac function in sepsis
Mitochondria and SICD | within 72 hours post admission
  examining the potential roles for increased reactive oxygen species (ROS) and nitric oxide (NO) production in SICD using mouse models of sepsis have shown that genetic and/or pharmacologic manipulation of these species decreased oxidative stress, increased ATP generation and restored cardiac function in sepsis
Mitochondria and SICD | after clinical recovery from sepsis (approximately 1 month)
  examining the potential roles for increased reactive oxygen species (ROS) and nitric oxide (NO) production in SICD using mouse models of sepsis have shown that genetic and/or pharmacologic manipulation of these species decreased oxidative stress, increased ATP generation and restored cardiac function in sepsis
Mitochondrial mechanisms to influence SICD | within 6 hours of admission to the ICU
  changes in mitochondrial bioenergetics associated with sepsis can result in differential releases of mtDNA DAMPs, which contribute in inflammation.
Mitochondrial mechanisms to influence SICD | within 72 hours post admission
  changes in mitochondrial bioenergetics associated with sepsis can result in differential releases of mtDNA DAMPs, which contribute in inflammation.
Mitochondrial mechanisms to influence SICD | after clinical recovery from sepsis (approximately 1 month)
  changes in mitochondrial bioenergetics associated with sepsis can result in differential releases of mtDNA DAMPs, which contribute in inflammation.
Mitochondrial bioenergetics and mtDNA DAMPs | within 6 hours of admission to the ICU
  determine the mitochondrial bioenergetic profiles from platelets isolated from blood samples collected from sepsis patients and controls.
Mitochondrial bioenergetics and mtDNA DAMPs | within 72 hours post admission
  determine the mitochondrial bioenergetic profiles from platelets isolated from blood samples collected from sepsis patients and controls.
Mitochondrial bioenergetics and mtDNA DAMPs | after clinical recovery from sepsis (approximately 1 month)
  determine the mitochondrial bioenergetic profiles from platelets isolated from blood samples collected from sepsis patients and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Riaz Karukappadath, MD, Principal Investigator — Department of Anesthesiology and Perioperative Medicine, Division of Critical Care Medicine
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined